CLINICAL TRIAL: NCT03919123
Title: Evaluation of Functional Outcomes and Quality of Life After Laparoscopic Promontofixation (PFL). Unicentric Retrospective Cohort Study (PeSuLife)
Brief Title: Evaluation of Functional Outcomes After Laparoscopic Promontofixation (PFL).
Acronym: PeSuLife
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A02927-48
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Pelvic Organ Prolapse; Symptoms; Satisfaction; Quality of Life
Keywords: Pelvic Organ Prolapse; laparoscopic promontofixation; symptoms; Satisfaction; Quality of Life
MeSH Terms: conditions — Pelvic Organ Prolapse; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation of laparoscopic promontofixation — Evaluation of Functional Outcomes and Quality of Life After Laparoscopic Promontofixation (PFL). Unicentric Retrospective Cohort Study (PeSuLife)

SUMMARY:
Prolapse of the pelvic organs is a common pathology in women with a strong impact on the quality of life. Its prevalence tends to increase due to increased life expectancy and obesity.

The main treatment is surgical and involves all organ specialists dealing with pelvic-perineal functional disorders: urologists, gynecologists, digestive surgeons.

Our team wishes to evaluate, on a cohort of patients operated at the Caen University Hospital, the functional uro-gynecologic, digestive and sexual results of pelvic organ prolapse (POP) repair by Laparoscopic Promontofixation (PFL) through symptoms and quality of life validated questionnaires (QoL).

The analysis of the responses to these questionnaires will allow us to evaluate the functional results in the short and medium term (from 6 months to 5 years)

DETAILED DESCRIPTION:
This is a retrospective cohort study conducted at the Universitary hospital of Caen in three surgical departments (gynecology, urology and digestive surgery).

Patients who had a laparoscopic promontofixation will be asked to respond to validated questionnaires of symptoms and quality of life after their surgery (PFDI-20, ICIQ-SF, PFIQ-7) and satisfaction (PGI-I)

ELIGIBILITY:
Inclusion Criteria:

Patients who have had a laparoscopic promotofixation for genital prolapse at the University Hospital of Caen between 2013 and 2018 in the departments of gynecology, urology and digestive surgery.

Patient who received written information and agreed to participate in the study

Exclusion Criteria:

Minor patient, under guardianship, under trusteeship Patient not understanding French Refusal to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 18 years old who underwent a laparoscopic promontofixation for pelvic organ prolapse at the University Hospital of Caen between 2013 and 2018 in the departments of gynecology, urology and digestive surgery, and agreed to participate in the study after a written information
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Effect of laparoscopic promontofixation on urogynecologic and digestive symptoms | 3 years
  The main objective is to collect the PFDI-20 score after the surgery. This score was developped to evaluate the genital, anorectal and digestive symptoms related to prolapse

SECONDARY OUTCOMES:
Effect of laparoscopic promontofixation on urinary incontinence | 3 years
  Assessment of the ICIQ-SF score, a specific score developped to assess the impact urinary incontinence
Sexual impact of laparoscopic promontofixation | 3 years
  Evaluation of the PISQ-12 score after laparoscopic promontofixation. This score was developped specifically to evaluate sexual troubles in case of genital prolapse
Evaluation of quality of life after prolapse surgery | 3 years
  Evaluation of the quality of life using a score specifically developped in case of genital prolapse : the PFIQ-7 score
Assessment of patient satisfaction after surgery | 3 years
  Evaluation of the quality of life using the PGI-I score, developped to quantify the effect of urinary or prolapse treatments
Specific evaluation of functional outcomes of laparoscopic rectopexy in rectocele or elytrocele indications | 3 years
  Evaluation of the PFDI-20 score in women undergoing laparoscopic rectopexy
Comparison of the different scores according to the operative indication (anterior promontofixation, double promontofixation, rectopexy alone) | 3 years
  Comparison of the PFDI-20 scores according to the operative indication

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Cécile Pizzoferrato, MD, PhD, Study Director — Universitary hospital of Caen
Locations (1):
- University Hospital, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fritel X, Varnoux N, Zins M, Breart G, Ringa V. Symptomatic pelvic organ prolapse at midlife, quality of life, and risk factors. Obstet Gynecol. 2009 Mar;113(3):609-616. doi: 10.1097/AOG.0b013e3181985312. PMID 19300324
- [Background] Lousquy R, Costa P, Delmas V, Haab F. [Update on the epidemiology of genital prolapse]. Prog Urol. 2009 Dec;19(13):907-15. doi: 10.1016/j.purol.2009.09.011. Epub 2009 Nov 4. French. PMID 19969258
- [Background] Adjoussou SA, Bohoussou E, Bastide S, Letouzey V, Fatton B, de Tayrac R. [Functional symptoms and associations of women with genital prolapse]. Prog Urol. 2014 Jun;24(8):511-7. doi: 10.1016/j.purol.2013.11.015. Epub 2013 Dec 27. French. PMID 24875570
- [Background] Le Normand L, Cosson M, Cour F, Deffieux X, Donon L, Ferry P, Fatton B, Hermieu JF, Marret H, Meurette G, Cortesse A, Wagner L, Fritel X. Clinical Practice Guidelines: Synthesis of the guidelines for the surgical treatment of primary pelvic organ prolapse in women by the AFU, CNGOF, SIFUD-PP, SNFCP, and SCGP. J Gynecol Obstet Hum Reprod. 2017 May;46(5):387-391. doi: 10.1016/j.jogoh.2017.05.001. Epub 2017 May 12. No abstract available. PMID 28506877
- [Background] Maher C, Feiner B, Baessler K, Schmid C. Surgical management of pelvic organ prolapse in women. Cochrane Database Syst Rev. 2013 Apr 30;(4):CD004014. doi: 10.1002/14651858.CD004014.pub5. PMID 23633316
- [Background] Maher CF, Feiner B, DeCuyper EM, Nichlos CJ, Hickey KV, O'Rourke P. Laparoscopic sacral colpopexy versus total vaginal mesh for vaginal vault prolapse: a randomized trial. Am J Obstet Gynecol. 2011 Apr;204(4):360.e1-7. doi: 10.1016/j.ajog.2010.11.016. PMID 21306698
- [Background] Lucot JP, Cosson M, Bader G, Debodinance P, Akladios C, Salet-Lizee D, Delporte P, Savary D, Ferry P, Deffieux X, Campagne-Loiseau S, de Tayrac R, Blanc S, Fournet S, Wattiez A, Villet R, Ravit M, Jacquetin B, Fritel X, Fauconnier A. Safety of Vaginal Mesh Surgery Versus Laparoscopic Mesh Sacropexy for Cystocele Repair: Results of the Prosthetic Pelvic Floor Repair Randomized Controlled Trial. Eur Urol. 2018 Aug;74(2):167-176. doi: 10.1016/j.eururo.2018.01.044. Epub 2018 Feb 19. PMID 29472143
- [Background] Paraiso MF, Walters MD, Rackley RR, Melek S, Hugney C. Laparoscopic and abdominal sacral colpopexies: a comparative cohort study. Am J Obstet Gynecol. 2005 May;192(5):1752-8. doi: 10.1016/j.ajog.2004.11.051. PMID 15902189
- [Background] Hsiao KC, Latchamsetty K, Govier FE, Kozlowski P, Kobashi KC. Comparison of laparoscopic and abdominal sacrocolpopexy for the treatment of vaginal vault prolapse. J Endourol. 2007 Aug;21(8):926-30. doi: 10.1089/end.2006.0381. PMID 17867956
- [Background] Ganatra AM, Rozet F, Sanchez-Salas R, Barret E, Galiano M, Cathelineau X, Vallancien G. The current status of laparoscopic sacrocolpopexy: a review. Eur Urol. 2009 May;55(5):1089-103. doi: 10.1016/j.eururo.2009.01.048. Epub 2009 Feb 4. PMID 19201521
- [Background] Chevrot A, Droupy S, Linares E, de Tayrac R, Costa P, Wagner L. [Impact of laparoscopic sacrocolpopexy on symptoms, health-related quality of life and sexuality: A 3-year prospective study]. Prog Urol. 2016 Sep;26(10):558-65. doi: 10.1016/j.purol.2016.02.009. Epub 2016 Mar 24. French. PMID 27052819
- [Background] Loffeld CJ, Thijs S, Mol BW, Bongers MY, Roovers JP. Laparoscopic sacrocolpopexy: a comparison of Prolene and Tutoplast mesh. Acta Obstet Gynecol Scand. 2009;88(7):826-30. doi: 10.1080/00016340902883158. PMID 19353330
- [Background] Deprest J, De Ridder D, Roovers JP, Werbrouck E, Coremans G, Claerhout F. Medium term outcome of laparoscopic sacrocolpopexy with xenografts compared to synthetic grafts. J Urol. 2009 Nov;182(5):2362-8. doi: 10.1016/j.juro.2009.07.043. Epub 2009 Sep 16. PMID 19762041
- [Background] Govier FE, Kobashi KC, Kuznetsov DD, Comiter C, Jones P, Dakil SE, James R Jr. Complications of transvaginal silicone-coated polyester synthetic mesh sling. Urology. 2005 Oct;66(4):741-5. doi: 10.1016/j.urology.2005.04.027. PMID 16230128
- [Background] Sergent F, Resch B, Loisel C, Bisson V, Schaal JP, Marpeau L. Mid-term outcome of laparoscopic sacrocolpopexy with anterior and posterior polyester mesh for treatment of genito-urinary prolapse. Eur J Obstet Gynecol Reprod Biol. 2011 Jun;156(2):217-22. doi: 10.1016/j.ejogrb.2011.01.022. Epub 2011 Feb 26. PMID 21353736
- [Background] Antiphon P, Elard S, Benyoussef A, Fofana M, Yiou R, Gettman M, Hoznek A, Vordos D, Chopin DK, Abbou CC. Laparoscopic promontory sacral colpopexy: is the posterior, recto-vaginal, mesh mandatory? Eur Urol. 2004 May;45(5):655-61. doi: 10.1016/j.eururo.2004.01.004. PMID 15082210
- [Background] D'Hoore A, Penninckx F. Laparoscopic ventral recto(colpo)pexy for rectal prolapse: surgical technique and outcome for 109 patients. Surg Endosc. 2006 Dec;20(12):1919-23. doi: 10.1007/s00464-005-0485-y. PMID 17031741
- [Background] Barber MD, Kuchibhatla MN, Pieper CF, Bump RC. Psychometric evaluation of 2 comprehensive condition-specific quality of life instruments for women with pelvic floor disorders. Am J Obstet Gynecol. 2001 Dec;185(6):1388-95. doi: 10.1067/mob.2001.118659. PMID 11744914
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Srikrishna S, Robinson D, Cardozo L. Validation of the Patient Global Impression of Improvement (PGI-I) for urogenital prolapse. Int Urogynecol J. 2010 May;21(5):523-8. doi: 10.1007/s00192-009-1069-5. Epub 2009 Dec 15. PMID 20013110